CLINICAL TRIAL: NCT06637267
Title: Prospective Evaluation of Proclarix® Test to Improve Risk Stratification in Men Scheduled for MpMRI and Prostate Biopsy in Cantonal Hospital Aarau
Status: Recruiting | Type: Observational
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, PD Dr. med. Maciej Kwiatkowski, PD Dr. med. Maciej Kwiatkowski, Senior Consultant with a Special Function, Head of Clinical Research Urology, Kantonsspital Aarau
Other Study IDs: 00175
Record Dates: First submitted 2024-10-02; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
Keywords: Proclarix
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection and storage of 40 ml serum to measure the Proclarix biomarkers ( Thrombospondin 1 (THBS1) and Cathepsin D (CTSD)as well as %fPSA and tPSA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Proclarix® — The aim of the study is the implementation of new biomarkers (Proclarix®) in order to increase the sensitivity and specificity of PSA-based Prostate cancer early detection avoiding unnecessary prostate biopsies thus decreasing the associated morbidity (infections, bleeding, urinary retention, etc.). PSA values, Proclarix and mpMRI findings will be correlated with the results of the prostate biopsy in order to improve patient selection for future biopsies in order to avoid unnecessary prostate biopsies, but still be able to detect relevant carcinomas at an early stage. The null hypothesis in our observational study is the lack of superiority in PCa early detection when using the Proclarix over PSA alone.
  Other Names: Proclarix risk score

SUMMARY:
The use of prostate-specific antigen (PSA) for the screening of prostate cancer has led to higher detection rates and a shift to lower and therefore potentially more curative disease stages at diagnosis and thus subsequently to a lower mortality. A suspicious digital rectal examination of the prostate or an increased PSA value are suspicious for PCa and indicate a confirmatory prostate biopsy . Almost 25% of all men report moderate to severe pain after the biopsy. Serious complications such as urosepsis requiring intensive medical monitoring are less common. There are also other predictors for the presence of prostate cancer: including positive family history in first-degree relatives, low PSA-ratio (= ratio between free to total PSA), older age and African-American race. In order to reduce the number of unnecessary prostate biopsies, numerous prostate-cancer risk calculators based on these predictors have been designed. Risk-calculators serve as an aid to clinical decision-making. For example, if the calculated risk of prostate cancer is low, a PSA follow-up can be a viable alternative to prostate biopsy. However, these risk calculators often have some shortcomings. The two most frequently used calculators are based on cohorts of men in whom the biopsies were performed as part of a study protocol regardless of the clinical context. These cohorts do not realistically represent the collective of patients to whom a prostate biopsy is indicated. Furthermore, the cohorts of these calculators are mostly very old and do not take into account the technical developments with improved sensitivity/specificity in recent years. Nowadays, a multiparametric magnetic resonance imaging (mpMRI) of the prostate is being performed and suspicious areas in the prostate are explicitly targeted, leading to an improved detection of significant carcinoma.The possibility of determining novel laboratory predictors such as biomarkers has been lately under investigation. All of these biomarkers are not included in the currently available risk calculators or are poorly validated. A pathological grading system, the so-called Gleason score, is a pathological grading system differentiating between less versus more aggressive prostate cancer cells. The most frequently used risk calculators have been developed based on patient cohorts that were created at a time before the Gleason score was revised to its current status. Thus, many previously low-grade carcinomas would be classified as more aggressive ones according to current pathology guidelines. Based on these circumstances, the development of a new PCa risk stratification models is of major clinical importance. In addition, as all biomarker measurements rely heavily on analytical performance of laboratory equipment, the quality assurance is an important factor and should be under scrutiny, especially when new biomarkers are under investigation.

Proclarix is a CE-marked test based on two new biomarkers, Thrombospondin 1 (THBS1) and Cathepsin D (CTSD), combined with PSA values and the patient's age. A software algorithm returns a risk assessment that can be utilized to predict clinically significant PCa (ISUP group 2 or higher).

DETAILED DESCRIPTION:
Hypothesis and primary objective The aim of the study is the implementation of new biomarkers (Proclarix) in order to increase the sensitivity and specificity of PSA-based PCa early detection avoiding unnecessary prostate biopsies thus decreasing the associated morbidity (infections, bleeding, urinary retention, etc.). PSA values, Proclarix and mpMRI findings will be correlated with the results of the prostate biopsy in order to improve patient selection for future biopsies in order to avoid unnecessary prostate biopsies, but still be able to detect relevant carcinomas at an early stage. The null hypothesis in our observational study is the lack of superiority in PCa early detection when using the Proclarix over PSA alone.

Primary and secondary endpoints The primary endpoint is the sensitivity and specificity of the Proclarix risk score in relation to the prediction of significant prostate cancer (Gleason score >7) in the prostate biopsy. These parameters should be compared to PSA, %fPSA and the mpMRI findings.

The secondary endpoints:

The correlation of the data collected from mpMRI (according to PI-RADS) to the biopsy results. The combination of clinical parameters, PSA values, Proclarix, mpMRI and pathology results in order to develop predictive risk stratification tool (e.g. risk score or nomogram) for PCa.

Determination of the analytical performance of the recently introduced Alinity i-Systems for PSA determination compared to the Architect i2000sr system (Abbott Laboratories) in terms of precision and validation of the reference interval according to the CLSI guidelines.

The study design of this single-center, single-arm, non-blinded prospective study includes the collection and storage of 40 ml serum from all patients who meet the inclusion criteria according to point 3.1 and are planned for a prostate biopsy as part of the routine clinical PCa workup with mpMRI of the prostate starting from September 2021. While participants are going to be recruited in prospective manner and asked for their consent, the Proclarix biomarkers as well as %fPSA and tPSA will be determined post-interventionally (analog to the PROPOSE trial).

According to the power analysis, 480 samples are necessary to achieve a 25%, statistically significant improvement in the negative predictive value of Proclarix compared to MPSA, assuming that 50% or more of all patients have a positive biopsy.

The mpMRI findings and biopsy results should be analyzed by frequency distribution and compared by standard statistical testing.The design of a risk stratification tool should be achieved by means of logistic regression analysis. Various parameter combinations should be compared by standard statistical testing.In order to evaluate the performance of the recently introduced Alinity i system for PSA assays in terms of precision and correlation compared to the Architect i2000sr system (Abbott Laboratories) and to validate the reference interval according to CLSI guidelines, approximately 100 serum samples will be included for the comparison of the two methods by means of standard statistical testing. SPSS v.24 standard statistical package will be used for the most of the data analysis. The statistical analysis will be performed with assistance of external statistician. P-value <0.05 or diverging boundaries of 95% confidence intervals will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Male patients between 45 and 80 years of age who are scheduled for an mpMRI followed by prostate biopsy (systematic and / or TRUS fusion biopsy) - within the framework of standard of care
* Signed ICE

Exclusion Criteria:

* patients who had previous treatments of the prostate (TUR prostate, cryoablation, HIFU, IRE, radiation therapy, alcohol instillation, etc.) in the past 5 years.
* acute urinary tract infections.
* the use of 5-alpha reductase inhibitors.
* mpMRI performed outside of the scope of Kantonsspital Aarau.

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients
Study Population: Male patients between 45 and 80 years of age who are scheduled for an mpMRI followed by prostate biopsy (systematic and / or TRUS fusion biopsy) - within the framework of standard of care
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the Proclarix risk score detenging clinically relevant prostate cancer. | August 2022 - July 2024
  The primary endpoint is the sensitivity and specificity of the Proclarix risk score in relation to the prediction of significant prostate cancer (Gleason score >7) in the prostate biopsy. These parameters should be compared to PSA, %fPSA and the mpMRI findings.

SECONDARY OUTCOMES:
The correlation of the data collected from mpMRI (according to PI-RADS) to the biopsy results. | August 2022 - July 2024
  The correlation of the data collected from mpMRI (according to PI-RADS) to the biopsy results.
The combination of clinical parameters, PSA values, Proclarix, mpMRI and pathology results in order to develop predictive risk stratification tool (e.g. risk score or nomogram) for PCa. | August 2022 - July 2024
  The combination of clinical parameters, PSA values, Proclarix, mpMRI and pathology results in order to develop predictive risk stratification tool (e.g. risk score or nomogram) for PCa.
Development of a Predictive Risk Stratification Tool for Clinically Significant Prostate Cancer | August 2022 to December 2025
  This outcome measure focuses on the development of a predictive risk stratification tool for identifying clinically significant prostate cancer (Gleason score ≥7). The tool will combine multiple clinical and diagnostic parameters, including:
  * Prostate-Specific Antigen (PSA) levels measured in ng/mL.
  * Multiparametric MRI (mpMRI) findings, assessed using the PI-RADS score (Prostate Imaging Reporting and Data System).
  * Proclarix risk score, a biomarker-based tool for prostate cancer risk assessment.
  * Pathology results from prostate biopsy, specifically Gleason scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Cantonal Hospital Aarau, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Results will be published by the investigators in academic journals. Sharing of generated study data will be carried out in several different ways. The investigator plan to make our results available to researchers and potential collaborators interested in prostate cancer screening